CLINICAL TRIAL: NCT05156788
Title: A Single-arm, Multi-center, Phase II Study of Tislelizumab, Lenvatinib and GEMOX Transformation in the Treatment of Potentially Resectable, Locally Advanced Biliary Tract Cancer
Brief Title: Tislelizumab（Anti PD-1), Lenvatinib and GEMOX Transformation in the Treatment of Potentially Resectable, Locally Advanced Biliary Tract Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZSAB-TransGOLP
Record Dates: First submitted 2021-09-30; First posted 2021-12-14 (Actual); Last update posted 2023-08-15 (Actual); Status verified 2023-08

CONDITIONS: Biliary Tract Cancer; PD-1 Antibody; Gemox; Lenvatinib
MeSH Terms: conditions — Biliary Tract Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PD-1 antibody +Lenvatinib+Gemox (Experimental): Tilelizumab 200mg, d1 Q3W Lenvatinib 8mg, po, qd, Gemox chemotherapy Gemcitabine 1000mg/m2, d1, 8, Q3W, + oxaliplatin 85mg/m2 d1, Q3W
  Interventions: Drug: PD-1+Lenvatinib+GEMOX

INTERVENTIONS:
Drug: PD-1+Lenvatinib+GEMOX — Tilelizumab 200mg, add 0.9% NS 100mL, d1 Q3W, Lenvatinib 8mg, po, qd Gemox chemotherapy: Gemcitabine 1000mg/m2 with 0.9% NS 100mL, 30 minutes, d1, 8, Q3W, + oxaliplatin 85mg/m2 with 5%GS 500mL, 2 hours, d1, Q3W

SUMMARY:
The aim of this study is to assess the R0 resection rate of tislelizumab combined with Lenvatinib and Gemox chemotherapy in the conversion therapy of potentially resectable locally advanced BTC.

DETAILED DESCRIPTION:
Translational therapy refers to methods such as chemotherapy, radiotherapy, immunotherapy, targeted and combined therapy to shrink tumors, reduce tumor biological behavior, and achieve secondary resection. The success rate of transformation depends on the objective response rate of the treatment method (Objective response rate, ORR). The latest review showed that 132 patients with unresectable ICC had undergone chemotherapy, chemoembolization, radiotherapy embolization or combination therapy, and 27 patients received downgrade resection. The research of our group using PD-1 antibody combined with lenvatinib and Gemox chemotherapy in the first-line treatment of unresectable advanced cholangiocarcinoma (NCT03951597, 2020ESMO, 2021ASCO) showed that the ORR was 80% and the disease control rate (DCR) It reached 93.3% (28/30), of which 3 cases underwent successful radical resection after downstage. These data suggest that PD1 monoclonal antibody combined with lenvatinib and Gemox chemotherapy may be an ideal conversion therapy for patients with potentially resectable advanced biliary system tumors, but there is currently no evidence-based basis.

This study explores the efficacy and safety of PD1 monoclonal antibody combined with Lenvatinib and Gemox chemotherapy in potentially resectable advanced BTC conversion therapy. It has certain clinical significance in order to increase the R0 surgical resection rate of BTC patients and improve patient survival.

ELIGIBILITY:
Inclusion Criteria:

* 1. Male or female aged 18-70 2. The patient must sign an informed consent form before joining the group, understand and be willing to sign a written informed consent form 3. Potentially resectable locally advanced BTC (including ICC, PBDT and GBC) confirmed by histology or cytology, agree to provide previously stored tumor tissue specimens or fresh biopsy tumor lesions for biomarker detection 4. Local progress, failure to achieve R0 resection, and no distant metastasis, with potential resection 5. At least one measurable lesion (RECIST 1.1) 6. Have never received systemic treatment for biliary tumors in the past 7. Eastern Cooperative Oncology Group (ECOG) performance status score ECOG PS 0-1 8. Liver function classification is Child-Pugh A 9. The bone marrow, liver and kidneys are fully functional and reach the following clinical laboratory evaluation standards within 7 days before treatment:

Blood indicators:

Absolute neutrophil count (ANC) ≥ 1.5 × 109/L, platelet ≥ 90 × 109/L, hemoglobin ≥ 90 g/L.

Liver function indicators:

AST and ALT are both ≤3×ULN (upper limit of normal value); total bilirubin ≤1.5×ULN

Kidney function indicators:

Serum creatinine≤1.5×ULN

Coagulation index:

International normalized ratio (INR) ≤ 1.2 or prothrombin time (PT) ≤ 1.2×ULN

Obstructive jaundice, after PTCD or ERCP treatment, if the liver function indicators meet the requirements for entry, it can be considered for entry:

10. If the subject has HBV or HCV infection, the following conditions must be met:

For inactive/asymptomatic carriers of HBV, chronic, or active HBV:

HBV deoxyribonucleic acid (DNA) <2000 copies/mL during the screening period. Remarks: Patients with HBV DNA>2000 copies/mL should be treated according to treatment guidelines. Patients who received antiviral drug treatment at the time of screening should have HBV-DNA <2000 copies/mL and continue treatment during the study period.

For subjects infected with HCV:

If the infection is confirmed based on the detectable HCV ribonucleic acid RNA, such subjects cannot be included in the group.

11. If you are a fertile woman (that is, physically capable of getting pregnant), you must agree to take effective contraceptive measures during the study period and within 120 days after the last administration, and have urine within 7 days before the first study drug administration Or the serum pregnancy test is negative.

12. If you are a non-sterilized male, you need to agree to take effective contraceptive measures during the study period and 120 days after the last dose.

13. Life expectancy ≥ 3 months

Exclusion Criteria:

* 1. Diagnosed as mixed type of periampullary carcinoma, hepatocellular carcinoma and cholangiocarcinoma 2. Have received systemic treatment for biliary tumors in the past 3. Have previously received gemcitabine-based chemotherapy or TKI therapy or any tumor immunotherapy (for example, PD-1/L1 inhibitors, CTLA-4 inhibitors, etc.) 4. Have a history of severe hypersensitivity to other monoclonal antibodies 5. Allergy to tislelizumab or any of its excipients; allergy to oxaliplatin and any of its excipients; allergy to gemcitabine and any of its excipients; allergy to lenvatinib and any of its excipients 6. The presence of pericardial effusion, uncontrollable pleural effusion or clinically obvious ascites within 7 days before treatment is defined as meeting the following criteria: (a) Ascites can be detected by physical examination during screening, or (b) during screening, Ascites requires puncture fluid.

  7. There is no clinical evidence of portal hypertension with esophageal or gastric varices within 6 months before starting treatment.

  8. Any bleeding or thrombotic disease or any anticoagulant (such as warfarin or similar drugs) that needs to monitor the international standardized ratio during treatment within 6 months before the start of treatment 9. Has suffered from any malignant tumors, except for the BTC studied in this clinical trial and locally recurring cancers that have been cured (such as resected basal cell or squamous cell skin cancer, superficial bladder cancer, cervical or breast cancer) Carcinoma in situ, occult carcinoma of the thyroid).

  10. Any known central nervous system metastasis and/or leptomeningeal disease have been present before treatment.

  11. A history of any active immunodeficiency or autoimmune disease and/or any immunodeficiency or autoimmune disease that may recur at the time of screening

Note: Subjects with the following diseases can be selected:

Type I diabetes Hypothyroidism (if only hormone replacement therapy can be used to control) Controlled celiac disease Skin diseases that do not require systemic treatment (eg vitiligo, psoriasis, hair loss) Any other disease that will not recur without external triggers 12. Any disease requiring systemic treatment with corticosteroids (dose higher than 10mg/day of prednisone or equivalent doses of similar drugs) or other immunosuppressive agents in the 14 days before treatment.

Remarks: Subjects who have currently or previously used any of the following steroid regimens can be selected:

In the absence of active autoimmune diseases, adrenaline replacement steroids are allowed (prednisone ≤10mg/day or equivalent dose of similar drugs) Local, ophthalmic, intra-articular, intranasal and inhaled corticosteroids with minimal systemic absorption Prophylactic short-term use (≤7 days) corticosteroids (for example, allergy to contrast agents) or for the treatment of non-autoimmune conditions (for example, delayed hypersensitivity reactions caused by contact allergens) 13. There is a history of interstitial lung disease or non-infectious pneumonia.

14. Any serious chronic infection or active infection (excluding viral hepatitis) that requires systemic antibacterial, antifungal or antiviral therapy (such as tuberculosis) before starting treatment.

15. The electrocardiogram during screening showed that the QT interval (QTc) corrected according to the heart rate (corrected according to the Fridericia method) exceeded 450 msec.

Note: If any patient finds that the QTc interval exceeds 450 msec during the first ECG examination, the ECG will be repeated to confirm the result.

16. Any of the following cardiovascular risk factors: Cardiogenic chest pain in the 28 days before treatment, defined as moderate pain that restricts daily activities (ADL) Symptomatic pulmonary embolism occurred within 28 days before treatment A history of acute myocardial infarction occurred within 6 months before treatment.

Any history of heart failure reaching New York Heart Association grade III or IV within 6 months of treatment Ventricular arrhythmia of grade ≥2 occurred within 6 months before treatment Cerebrovascular accident (CVA) or transient ischemic attack (TIA) occurred within 6 months before treatment.

17. Have received organ transplantation or hematopoietic stem cell transplantation (HSCT) or any major surgery within 28 days before treatment.

18. Known mental or substance abuse disorders that may interfere with test compliance.

19. Live vaccine has been vaccinated 28 days before treatment. Note: Seasonal influenza vaccines are generally inactivated influenza vaccines and are allowed to be used.

20. Known history of human immunodeficiency virus infection (HIV) or syphilis infection.

21. The history or evidence of any disease, treatment, or laboratory abnormality that may confuse the test results, interfere with the participation of the subject during the entire trial, or the main investigator believes that it does not meet the subject's best benefit.

22. Currently participating in and receiving treatment, or participating in or participating in other drug or device research within 4 weeks after the first administration of the research drug.

23. From the screening visit to 120 days after the last drug administration, pregnancy or breastfeeding, or expectation of pregnancy or childbirth within the planned duration of the trial.

24. The investigator judges that the compliance is not good, or there are other conditions that make the patients unsuitable to participate in this trial.

25. There are various medical contraindications that prevent the use of enhanced imaging (CT or MRI).

26. There are surgical contraindications, and the researchers believe that it is not suitable for surgical patients.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-12-12 (Actual); Primary Completion 2023-07-03 (Actual); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
R0 resection rate | 24 months
  the ratio of the number of R0 resection cases to the total number of enrolled cases

SECONDARY OUTCOMES:
ORR | 24 months
  The proportion of patients whose best overall response (BOR) is evaluated as achieving complete response (CR) or partial response (PR) at any time during study drug treatment
DCR | 24 months
  Proportion of patients with CR, PR and SD
PFS | 24 months
  Time from study treatment to disease progression or all-cause death as assessed by the investigator (whichever occurs first)
OS | 24 months
  The time from study treatment to the date of death of the subject, regardless of the cause of death
CPR | 24 months
  The ratio of the number of pathological complete necrosis of excised specimens to the total number of surgical resections
MPR | 24 months
  The ratio of more than 90% cases of pathological necrosis of resected specimens to the total number of surgical resections
RFS | 24 months
  Proportion of patients without tumor recurrence or metastasis after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Jia Fan, Principal Investigator — Shanghai Zhongshan Hospital
Locations (2):
- China (2):
  - Zhongshan hospital, Shanghai
  - Shenzhen University General Hospital, Shenzhen

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Shi G, Huang X, Li X, Liang F, Gao Q, Zhang D, Lu J, Ji Y, Hu Z, Chen Y, Qiu S, Yi Y, Zhu X, Sun H, Shi Y, Peng M, Wang X, Huang C, Ding Z, He Y, Shen Y, Xu Y, Xiao Y, Hu J, Zhou J, Fan J. Conversion therapy of tislelizumab plus lenvatinib and GEMOX in unresectable locally advanced biliary tract cancer (ZSAB-TransGOLP): a multicentre, prospective, phase 2 study. Lancet Oncol. 2025 Oct;26(10):1334-1345. doi: 10.1016/S1470-2045(25)00376-6. Epub 2025 Aug 29. PMID 40889502